CLINICAL TRIAL: NCT01475474
Title: A Multi-Center, Prospective, Non-Randomized Study of the Renew Insert Efficacy, Safety and Tolerability For the Management of Accidental Bowel Leakage Due to Bowel Incontinence
Brief Title: A Study to Evaluate the Safety, Tolerability and Effectiveness of the Renew Insert in Treating Accidental Bowel Leakage
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renew Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Renew Medical - 210CLD
Record Dates: First submitted 2011-11-10; First posted 2011-11-21 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-09

CONDITIONS: Bowel Incontinence
Keywords: incontinence; bowel; movement; fecal; anal; diarrhea; stool; rectal; feces; uncontrolled; loose; leakage; rectum; BM; watery; urgent; flatulence; gas
MeSH Terms: conditions — Fecal Incontinence; Diarrhea; Flatulence; Mucopolysaccharidosis IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Renew Insert — The Renew Insert is indicated for the management of accidental bowel leakage due to bowel incontinence. The Renew Insert is designed for self-insertion to seal and help prevent the involuntary leakage of stool from the rectum.

SUMMARY:
The purpose of this study is to determine whether the use of the Renew Insert is effective, tolerable and safe in the treatment of accidental bowel leakage due to bowel incontinence.

DETAILED DESCRIPTION:
Prospective, open label, single-arm, non-randomized, multi-center study designed to evaluate the efficacy, safety and tolerability of the Renew Insert in moderate-to-severe bowel incontinence patients: Minimum Wexner score of 12 AND at least weekly (score 3 or higher) leakage of solid and or liquid type stool.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Minimum Wexner Bowel incontinence score of 12 AND at least weekly (score of 3 or higher) leakage of solid and/or liquid type stool, with no greater than 50% of subjects with daily (score 4) of uncontrolled gas.
* Patients colon surveillance must be in compliance with American Cancer Society colon screening guidelines. If patient is out of compliance, they may be scheduled for Colonoscopy.
* Patient comprehends study meaning & is capable of carrying out study duties
* Fluent in English

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) score of 4 or higher
* Spinal cord injury or other major neurological diagnosis
* Known immune deficiency state
* Significant cardiac arrhythmia
* Pregnant or Breastfeeding
* Inflammatory bowel disease
* Requirement of medication delivered by suppository
* Active perianal abscess or fistula
* Present rectal prolapse
* Third degree hemorrhoids
* Anal stricture
* History or rectal spasm
* Rectal surgery in past 6 months
* Unresolved Anismus
* Fecal impaction with overflow diarrhea
* Ileo-anal pouch
* Rectocele requiring surgery
* Allergy to silicone or one of its components
* Significant medical condition which interferes with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Wexner, MD, Principal Investigator — Cleveland Clinic Florida; Emily Lukacz, MD, Principal Investigator — University of California, San Diego, CA; Mark Segall, MD, Principal Investigator — The medical office of Mark Segall MD; Eric G Weiss, MD, Principal Investigator — Cleveland Clinic Florida
Locations (3):
- United States (3):
  - Dr. Segall, Los Gatos, California
  - UCSD Medical Center, San Diego, California
  - Cleveland Clinic Florida, Weston, Florida

REFERENCES:
- [Derived] Lukacz ES, Segall MM, Wexner SD. Evaluation of an Anal Insert Device for the Conservative Management of Fecal Incontinence. Dis Colon Rectum. 2015 Sep;58(9):892-8. doi: 10.1097/DCR.0000000000000427. PMID 26252852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three (3) clinical sites participated in the US pivotal trial, enrolling a total of ninety-seven subjects. The trial consisted of a 4-week baseline evaluation period, a 12-week treatment period and a 4-week return to baseline period. The study started in December 2009 and completed in December 2011.
Pre-assignment Details: Renew Medical conducted a multi-center, prospective, open label, single-arm, non-randomized pivotal study designed to establish the safety, effectiveness, and tolerability of the Renew Insert in subjects with moderate-to severe bowel incontinence (defined as having a Wexner score greater than 12).
Groups:
- Renew Insert for Management of Accidental Bowel Leakage: The Renew Insert is designed for self-insertion to seal and help prevent involuntary leakage of stool from the rectum. The Insert is designed for single use and consists of two components: a soft, easily deformable silicone insert and a flexible plastic fingertip applicator. After self insertion into the anal canal the Insert is expelled with voluntary bowel movement or if desired, manually removed by the user.
Period: Baseline Period - 4 Weeks
Arm/Group | Renew Insert for Management of Accidental Bowel Leakage
Started | 97
Completed | 91
Not Completed | 6
Not completed — Did not meet eligibility for treatment | 4
Not completed — Withdrawal by Subject | 2
Period: Treatment Period - 12 Weeks
Arm/Group | Renew Insert for Management of Accidental Bowel Leakage
Started | 91
Completed | 73
Not Completed | 18
Period: Return to Baseline Period - 4 Weeks
Arm/Group | Renew Insert for Management of Accidental Bowel Leakage
Started | 73
Completed | 71
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Renew Insert for Management of Accidental Bowel Leakage
Number analyzed (Participants) | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 97

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Effectiveness Endpoint: A Relative Percentage Change in Episodes of Accidental Bowel Leakage (ABL) Determined by Comparing Treatment Results to Pre-treatment Results From the Baseline Period as Measured by Daily Diary Recordings.
Description: This co-primary effectiveness endpoint was calculated as a relative percentage of the baseline Accidental Bowel Leakage (ABL) using the following equation: % reduction in ABL = 100*(baseline period ABL - treatment period ABL) / (baseline period ABL)
Time Frame: Reduction in accidental bowel leakage from Baseline (Weeks 1-4) through Treatment period (Weeks 5-16).
Population: Primary cohort for the effectiveness analyses was the Modified Intent-To-Treat cohort which included all subjects who completed at least one week of Insert use during the 12 week Treatment Period.
Measure: Median (Inter-Quartile Range); unit: percentage change
Groups:
- Modified Intent-To-Treat Cohort: Modified Intent-to-Treat cohort included all subjects who completed week one and up to week 12 during the 12-Week Treatment Period.
Arm/Group | Modified Intent-To-Treat Cohort
Number analyzed (Participants) | 85
percentage change | -81.8 [-91.7 to -60.3]
Statistical Analysis 1: Comparison: Modified Intent-To-Treat Cohort; Wilcoxon Signed-Rank Test used to evaluate median Percent Change-from-Baseline in ABL different from zero; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed-Rank Test

2. Primary Outcome: Co-primary Effectiveness Endpoint: A Relative Percentage Change in Wexner Score (or Bowel Incontinence) Severity by Comparing Post-treatment Wexner Scores to Pre-treatment (End of Baseline Period) Wexner Scores.
Description: The Wexner fecal incontinence scale takes into account five parameters that are scored on a scale from zero (absent) to four (daily) frequency of incontinence to gas, liquid, solid, use of pad, and quality of life. Full continence is a Wexner total of zero (0), whereas full incontinence is a Wexner total of 20.
  This co-primary effectiveness endpoint is the mean % reduction in Wexner score from the baseline period to the end of the treatment period, which was calculated according to the following equation: % reduction in Wexner = 100% (baseline period Wexner - end treatment period Wexner) / (baseline period Wexner).
Time Frame: Wexner score was calculated at the end of the Baseline period (Weeks 1-4) to the end of the 12-Week Treatment Period (week 16).
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage change
Groups:
- Modified Intent to Treat Cohort (MITT): Modified Intent-to-Treat cohort included all subjects who completed at least one week of Insert use during the 12 Week Treatment Period.
Arm/Group | Modified Intent to Treat Cohort (MITT)
Number analyzed (Participants) | 77
Percentage change | -29.4 [-46.2 to 13.3]
Statistical Analysis 1: Comparison: Modified Intent to Treat Cohort (MITT); Wilcoxon Signed-Rank Test used to evaluate median Percent Change-from-Baseline in Wexner score; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed-Rank Test

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all subjects who used a Renew Insert through the end of study.
Groups:
- Intent-to-treat (ITT) Cohort: Subjects who used the Renew Insert.
Arm/Group | Intent-to-treat (ITT) Cohort
Serious Adverse Events (participants affected / at risk) | 0/91
Other Adverse Events (participants affected / at risk) | 91/91
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intent-to-treat (ITT) Cohort (N=91)
Abdominal Pain (Gastrointestinal disorders) | 5
Accidental Bowel Leakage (Gastrointestinal disorders) | 5
Anorectal Bleeding (Gastrointestinal disorders) | 8
Anorectal Irritation (Gastrointestinal disorders) | 14
Anorectal Pain (Gastrointestinal disorders) | 6
Anorectal Soreness (Gastrointestinal disorders) | 12
Anorectal Urge (Gastrointestinal disorders) | 24
Diarrhea (Gastrointestinal disorders) | 11
Discomfort (Gastrointestinal disorders) | 5
Gas (Gastrointestinal disorders) | 5
Device Displacement (General disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other